CLINICAL TRIAL: NCT06004024
Title: Validity, Reliability, and Smallest Detectable Change of the Short Form 12-Item (SF-12) Health Survey in Individuals With Knee Osteoarthritis: A Cross-sectional Study
Brief Title: Psychometric Properties of the Short Form 12-item (SF-12) Health Questionnaire in Individuals With Knee Osteoarthritis
Acronym: SF-12
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meltem Meran Çağlar (Other)
Responsible Party: Sponsor-Investigator, Meltem Meran Çağlar, lecturer, Beykoz University
Organization: Beykoz University (Other)
Other Study IDs: MedipolU
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis; Quality of Life
Keywords: SF-12; knee osteoarthritis; validity; reliability; minimal detectable change
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Knee Osteoarthritis (OA) is one of the most common joint diseases with chronic low-severity inflammation. 80% of individuals with knee OA have limited movements; It was found that 25% of them could not do their daily work. In addition, it has been shown that the quality of life of individuals with OA is lower compared to healthy individuals. This showed that measuring and reporting quality of life should be mandatory in clinical studies conducted in individuals with knee OA. It was stated that the most frequently used general scales in the evaluation of quality of life in these individuals were SF-36 or SF-12. It takes a long time for the SF-36 to be filled by individuals, which creates a disadvantage for both patients and clinicians. Developed as a shorter alternative to SF-36, SF-12 has also been shown to give similar results to SF-36 in individuals with knee OA who have undergone total knee arthroplasty. However, the psychometric properties of SF-12 in individuals with knee OA have not been examined. The purpose of this study is to examine whether SF-12 is valid and reliable in individuals with knee OA and to determine the minimum detectable change (MDC) value.

DETAILED DESCRIPTION:
Forty volunteers aged 40 years and older diagnosed with knee OA will be included in the study. First, individuals will be informed about the study in detail, and signed informed consent form will be obtained from individuals who agree to participate in the study. First of all, the demographic information of the individuals will be recorded. Chronic diseases and continuous drug use will be questioned. Individuals' quality of life will be evaluated with the SF-12 and SF-36 scales, and their functional status will be evaluated with the WOMAC score. All scales will be filled once, but the second evaluation for the test-retest reliability (intra-rater reliability) of the SF-12 scale will be repeated one week later. In our study, the sample size was determined by using a web-based sample size calculation application specially developed for reliability-validity studies. In this application, hypothesis testing was performed according to ICC values. The minimum acceptable reliability (ICC) was 0.65 and the expected reliability from the study was 0.85. When the significance level of the study (α) was determined as 0.05 and the power of the study (1-β) was determined as 80%, and considering the probability that 10% of the individuals participating in the study could exit the study, it was found that the minimum sample size to be taken for the study should be 40 people. Jamovi 2.3.28 program will be used in the statistical analysis of the data. Variables determined by measurement will be expressed as mean ± standard deviation (X ± SD), percent (%) will be calculated for variables determined by counting. The normal distribution will be evaluated by examining both visually (Histogram and Q-Q plots) and statistical techniques (Kolmogorov Smirnov test, Skewness and Kurtosis values). Criterion-releated validity of SF-12 will be evaluated by its subtype, concurrent validity, and its correlation with WOMAC and SF-36 scales will be evaluated. Pearson correlation test will be applied when the correlation normal distribution conditions are met, and Spearman correlation test will be applied if not. Correlation coefficient level will be considered as <0.3 low, 0.3- 0.5 medium, >0.5 strong. In the reliability test of the SF-12 scale, test-re-test will be applied for the stability of the scale, and intra-class correlational coefficients (ICC) will be calculated. ICC values of 0.5-0.75 will indicate moderate reliability, 0.75-0.9 good reliability, and >0.9 excellent reliability. In order to determine the internal consistency of the scale, internal consistency coefficients (Cronbach's alpha) will be calculated. It will be at an acceptable level when Cronbach's alpha is >0.7. Absolute reliability will be determined by calculating the standard error of measurement (SEM) to ensure the accuracy of the measurement. The SEM will be used to calculate the smallest detectable change at the 95% confidence level (MDC95) and will be calculated as: MDC95=SEM × 1.95 × √2. In all statistics, the "p" significance value will be taken as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 40 years and older,
* Radiological and clinical diagnosis of knee OA,
* Volunteering to participate in the study,
* Ability to read and write

Exclusion Criteria:

* Having problems with cooperation or cognitive impairment,
* Previous total knee arthroplasty surgery,
* Presence of neurodegenerative or neuromuscular disease,
* Psychological disorders,
* Presence of depression

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research will be carried out in Aydın ARSLAN Orthopedics and Traumatology Clinic, which is connected to the province of Istanbul, in individuals aged 40 and over who are diagnosed with knee osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Health Status Questionnaire (Short Form-SF-36) | Evaluation data will be collected within six month.
  The SF-36 is a widely used self-reported general health status questionnaire that measures eight dimensions of health status. Physical functioning, role restrictions due to physical health problems, bodily pain, social functionality, general mental health, role restrictions due to emotional problems, vitality and general health perceptions. It is a form that evaluates the last 4 weeks. While these eight sub-dimensions can be scored separately, the physical and mental component summary score (FCS and MCS score, respectively; Physical and Mental Component Summary Scores) can be obtained by weighing them and providing a general assessment of physical and mental health.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Evaluation data will be collected within six month.
  WOMAC will be used to assess patients' knee pain, joint stiffness and function. WOMAC is a disease-specific health status measure frequently used in patients with knee and hip OA. WOMAC consists of 24 questions, 5 questions in the pain section, 2 questions in the stiffness section, and 17 questions in the function section.
Short Form 12-Item (SF-12) Health Survey | Evaluation data will be collected within six month.
  The 12-item short form health questionnaire (SF-12) is a measure of physical and mental health. It has been reported that SF-12, which was created from the original form, SF-36, is more advantageous in terms of ease of application and shorter completion time. While the PCS-12 score is obtained from the sub-dimensions of general health, physical functionality, physical role and body pain, the MCS-12 score is obtained from the sub-dimensions of social functionality, emotional role, mental health and energy.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Meran Çağlar, Study Chair — Medipol University
Locations (1):
- Meltem Meran Çağlar, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No